CLINICAL TRIAL: NCT06330051
Title: The Improve Acute Reperfusion Treatment Quality for Ischemic Stroke Through Spatiotemporal Computing in China (IMPROVE-II ) -A Multicenter, Evaluator-Blind, Cluster-Randomized Controlled Study
Brief Title: The Improve Acute Reperfusion Treatment Quality for Ischemic Stroke Through Spatiotemporal Computing in China
Acronym: IMPROVE-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zi-Xiao Li, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KY 2023-184-02
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
Keywords: ischemic stroke; intravenous thrombolysis; endovascular treatment; medical quality; spatiotemporal computing
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After 3 months of baseline information collection,20 hospitals will be randomly assigned to the control and intervention groups according to baseline DNT to reduce the imbalance between the two groups. We will not indicate to any hospital the grouping type of other hospitals. If the selected hospital is unable to complete the study for some reason during the operation, the hospital with conditions to carry out the replacement will be selected from the hospitals of the same region, the same level and the same scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Improvement intervention (Experimental): receive the following continuous improvement intervention for 8months
  Interventions: Behavioral: improvement acute reperfusion treatment quality for stroke through spatiotemporal computing
- Control group (No Intervention): Only information will be collected.

INTERVENTIONS:
Behavioral: improvement acute reperfusion treatment quality for stroke through spatiotemporal computing — 1. Intelligent bracelet automatic positioning device and data feedback system based on spatiotemporal computing technology
  2. Continuous in-hospital procedure improvement based on P-D-C-A cycle for AIS
  Arms: Improvement intervention

SUMMARY:
This study intends to construct the goal-oriented integrated intervention model for AIS in-hospital procedure through the spatiotemporal positioning and the P-D-C-A cycle for continuous improvement (FAST model). Then a multicenter, evaluator-blind, cluster-randomized controlled study aims to verify the validity and safety of this FAST model.

DETAILED DESCRIPTION:
This study intends to construct the goal-oriented integrated intervention model, namely the preset first aid of acute ischemic stroke (AIS) process is the key time node in the target, through the intelligent bracelet automatic positioning, feedback system with real-time data as the carrier, through the P (Plan)-D (Do)-C (Check)-A (Act) cycle for continuous improvement, so as to shorten the delay time of reperfusion therapy and improve the rate of intravenous thrombolysis in AIS patients.

Then a multicenter, evaluator-blind, cluster-randomized controlled study aims to verify the validity and safety of this FAST model. This study will recruit 20 secondary or tertiary hospitals that meet the inclusion criteria, mainly distributed in the Beijing-Tianjin-Hebei-Shanxi-Neimenggu region. After 3 months of baseline information collection, 20 hospitals will be randomly assigned to the control and intervention groups. Then, the intervention group will install intelligent bracelet automatic positioning device and data feedback system based on spatiotemporal computing for 4 months. As the knowledge gained from the training may affect the identification of AIS patients, the duration of the training will keep as short as possible. We will conduct training to ensure that only trained caregivers and researchers master the use of the application to maintain the integrity of the intervention. During this 4-month period, both the control group and the intervention group will cease data collection, entering a phase of silence in the study. The FAST model intervention based on spatiotemporal computing technology will uniformly start after installation and training in each intervention group hospital. The intervention group will receive continuous intervention with a goal-oriented integrated intervention model based the spatiotemporal computing technology for 8 months and collect information, mainly the critical time information of the AIS reperfusion therapy process. In the control group, only information will be collected.

We will compare the critical treatment time information, Door to Needle time and Door to Puncture time, etc., between the two groups and conduct a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Hospitals#

1. Secondary or tertiary public hospitals with an emergency department that receive patients with AIS.
2. Admit at least 50 patients of AIS within 4.5 hours after onset each month.
3. Have the capacity of intravenous thrombolytic therapy or/and endovascular treatment.
4. Voluntarily participate in this research and cooperate with the installation of bluetooth positioning device and the improvement of AIS emergency procedures.
5. Have good cooperation relationship among the department of Neurology, Emergency, Interventional department, Neurosurgery department, Laboratory department and Radiology department.
6. Have ability to establish or participate in the establishment of patient information database and arrange a person responsible for the collection of case information.

Patients# Patients who are ≥18 years old are eligible for inclusion if they present with AIS diagnosed by CT and/or MRI, arrive at hospital within 4.5 hours after symptom onset, sign the informed consent form and agree to follow up until 3 months after stroke onset.

Exclusion Criteria:

Hospitals#

1. Hospital that unable to cooperate and complete the research.
2. Hospitals that are participating in other AIS medical quality improvement projects or related clinical trials.

Patients#

1. Patients refuse to sign informed consent and follow up until 3 months after stroke onset.
2. Patients with mild nondisabling stroke symptoms (Defined as NIHSS≤3, as any of the following: isolated facial paralysis; mild cortical blindness; mild hemianesthesia; mild hemiataxia.)
3. Life expectancy three-months or less by judgment of the investigator.
4. Participation in any interventional study that may affect the outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-06-18 (Estimated); Study Completion 2025-09-18 (Estimated)

PRIMARY OUTCOMES:
The Door to Needle time (DNT) for intravenous thrombolytic therapy in eligible patients within 4.5 hours of onset. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.

SECONDARY OUTCOMES:
The Door to Puncture time (DPT) for endovascular treatment within 6 hours of onset in eligible patients admitted to hospital within 4.5 hours of onset. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
The rate of intravenous thrombolytic therapy in eligible patients within 4.5 hours of onset. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
The rate of endovascular treatment within 6 hours of onset in eligible patients admitted to hospital within 4.5 hours of onset. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Incidence of symptomatic intracranial hemorrhage (sICH) within 36 hours of receiving reperfusion therapy. | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
Proportion of patients with 90-day favorable functional outcome. | Participants will be followed for 3 month after stroke onset.
  mRS 0-1
Proportion of patients with 90-day independent functional outcome. | Participants will be followed for 3 month after stroke onset.
  mRS 0-2
in-hospital mortality | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
90-day mortality | Participants will be followed for 3 month after stroke onset.

CONTACTS AND LOCATIONS:
Locations (1):
- WuQing People's Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No